CLINICAL TRIAL: NCT02822820
Title: The Impact of Bipolar Energy Modalities on Peri-operative Outcome During Laparoscopic Staging Surgery of Gynecologic Cancers: A Randomized Clinical Trial
Brief Title: The Comparison of Conventional and Advanced Bipolar Energy Modalities During Laparoscopic Staging Surgery of Gynecologic Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, salih taskin, Assoc. Prof., Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03
Record Dates: First submitted 2016-06-24; First posted 2016-07-04 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Perioperative Period

ARMS (2):
- Advanced bipolar (Ligasure-Covidien) (Active Comparator): Devices with advanced bipolar energy (Ligasure-Covidien) will be used during laparoscopic hysterectomy and pelvic lymphadenectomy
  Interventions: Device: Ligasure-Covidien
- Conventional bipolar (RoBi forceps-Karl Storz) (Active Comparator): Devices with conventional bipolar energy (RoBi rotating bipolar forceps-Karl Storz) will be used during laparoscopic hysterectomy and pelvic lymphadenectomy
  Interventions: Device: RoBi forceps-Karl Storz

INTERVENTIONS:
Device: Ligasure-Covidien — Vessel sealing device Ligasure-Covidien used during laparoscopic hysterectomy and pelvic lymphadenectomy
  Arms: Advanced bipolar (Ligasure-Covidien)
Device: RoBi forceps-Karl Storz — Vessel sealing device RoBi forceps-Karl Storz used during laparoscopic hysterectomy and pelvic lymphadenectomy
  Arms: Conventional bipolar (RoBi forceps-Karl Storz)

SUMMARY:
This single-institution prospective randomized clinical trial will be performed at the Gynecologic Oncology clinic of Ankara University. Patients with endometrial cancer and cervix cancer who will be operated for staging via laparoscopic approach will be included in the study. The included patients will be randomized to two groups before surgery. During the operation of first group instruments with advanced bipolar energy will be used during lymphadenectomy and hysterectomy and salpingo-oophorectomy. In the second group the operation will be performed by conventional bipolar energy forceps. The outcome parameters to be measured are intra-operative bleeding, duration of operation, intraoperative complications, postoperative pain score, postoperative complications, postoperative duration of hospitalization, late complications such as lymphocele formation and costs.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of endometrial or cervix cancer
* Stage I, IB1, IIA1 cervix cancer or patients with partial or complete response to chemoradiotherapy
* Clinically stage I and II endometrial cancer

Exclusion Criteria:

* Hematologic abnormality
* Coagulation disorder
* Present or past thromboembolic disease
* ECOG performance >2
* Advanced stage disease
* Fertility preserving surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Duration of operation | six months
Perioperative complications | six months

SECONDARY OUTCOMES:
Pain measured by Visual Analog Scale | Postoperative pain scores at 8th and 24th hours
Total cost of hospitalization, operation and complications | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Medical Faculty Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Taskin S, Sukur YE, Altin D, Turgay B, Varli B, Baytas V, Ortac F. Bipolar Energy Instruments in Laparoscopic Uterine Cancer Surgery: A Randomized Study. J Laparoendosc Adv Surg Tech A. 2018 Jun;28(6):645-649. doi: 10.1089/lap.2017.0639. Epub 2018 Jan 11. PMID 29323616